CLINICAL TRIAL: NCT00552045
Title: Epilepsy Phenome/Genome Project: A Phenotype/Genotype Analysis of Epilepsy
Brief Title: Epilepsy Phenome/Genome Project
Acronym: EPGP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01NS053998-01A1; CRC; 1R01NS053998 (Other: This is an NIH grant number, but it will not accept it as one.)
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Epilepsy; Localization-related Epilepsy; Infantile Spasms; Lennox-Gastaut Syndrome; Polymicrogyria; Periventricular Heterotopias
Keywords: epilepsy; localization-related epilepsy; idiopathic generalized epilepsy; infantile spasms; Lennox-Gastaut syndrome; polymicrogyria; periventricular heterotopias; malformations of cortical development; phenome; genome; genotype; phenotype
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Spasms, Infantile; Lennox Gastaut Syndrome; Polymicrogyria; Periventricular Nodular Heterotopia; Epilepsy, Idiopathic Generalized; Malformations of Cortical Development

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- subject: individuals with epilepsy

SUMMARY:
The purpose of this study is to collect detailed information about the characteristics and genetics of a large number of individuals with epilepsy.

DETAILED DESCRIPTION:
Epilepsy is one of the most common neurological disorders and is a major public health concern. Approximately 30 percent of people with epilepsy have medically intractable epilepsy, and the medical and social consequences of the disorder are enormous. Treatments developed for epilepsy have largely been experimental rather than based on knowledge of basic mechanisms because the mechanisms are poorly understood.

The Epilepsy Phenome/Genome Project (EPGP) is a large-scale, international, multi-institutional, collaborative research project aimed at advancing the understanding of the genetic basis of the most common forms of epilepsy.

The overall goal of EPGP is to collect detailed, high quality phenotypic (i.e., characteristics of individuals, from the molecular level to the whole person) information on persons with epilepsy and to compare the phenotypic information with genomic information. EPGP will provide a resource that may lead to many discoveries related to the diagnosis and treatment of epilepsy, including the eventual development of new therapies based on a better understanding of causes of the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Current age from 4 weeks to 60 years.
* Clear diagnosis of epilepsy, i.e., a lifetime history of two or more unprovoked seizures.
* Age at first unprovoked seizure younger than 40 years.
* High quality clinical and laboratory data (i.e., neuroimaging, EEG) must be available throughout the patient's history
* All patients with localization-related epilepsy (LRE) or idiopathic generalized epilepsy (IGE) must have a first-degree relative (parent, child, or sibling) with non-symptomatic (idiopathic or cryptogenic) epilepsy who is willing and available to participate.
* All patients with infantile spasms (IS), Lennox-Gastaut syndrome (LGS), or malformations of cortical development (MCD) must have both biological parents available and willing to participate.

Exclusion Criteria:

* Clinical and laboratory data do not allow a clear determination of whether the patient has epilepsy, or whether the diagnosis is LRE, IGE, IS, LGS, or MCD.
* Exclusively febrile seizures or other acute symptomatic seizures.
* Identified antecedent cause of epilepsy (i.e., a structural or metabolic insult to the CNS prior to the first unprovoked seizure, such as stroke, brain tumor, severe head trauma, etc., or a progressive neurodegenerative disorder).
* Recognized genetic syndrome (e.g., tuberous sclerosis, neurofibromatosis, Rett's or Angelman's syndromes) or chromosomal abnormality. (e.g., aneuploidies, unbalanced translocations, or chromosomal deletions and duplications detectable by conventional medical karyotyping).

Ages: 4 Weeks to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: EPGP will recruit persons with specific forms of epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 4150 (Actual)
Dates: Start 2007-11; Primary Completion 2013-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
EPGP will recruit persons with specific forms of epilepsy. DNA will be isolated from participants' blood and genetic variants associated with common forms of epilepsy will be identified. | over 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lowenstein, MD, Principal Investigator — University of California, San Francisco, Department of Neurology; Ruben Kuzniecky, MD, Principal Investigator — New York University, Comprehensive Epilepsy Center
Locations (25):
- United States (23):
  - University of Alabama at Birmingham, Epilepsy Center, 1719 6th Ave S, CIRC, Ste 312, Birmingham, Alabama
  - Mayo Clinic College of Medicine Arizona, Phoenix, Arizona
  - University of California, San Francisco, 400 Parnassus, Room 847, San Francisco, California
  - The Children's Hospital, Denver, Colorado
  - Mayo Clinic College of Medicine Florida, Jacksonville, Florida
  - Rush Presbyterian St. Luke's Medical Center, 1653 West Congress Parkway, Chicago, Illinois
  - Johns Hopkins University, Meyer 2-147, 600 North Wolfe Street, Baltimore, Maryland
  - Children's Hospital Boston, 300 Longwood Ave., Boston, Massachusetts
  - University of Michigan Medical Center, Department of Neurology, 5021 BSRB, 109 Zina Pitcher Place, Ann Arbor, Michigan
  - Mayo Clinic College of Medicine, 200 First St., SW, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Saint Barnabas Medical Center, Institute of Neurology, 101 Old Short Hills Road, 4th Floor, Suite #415, West Orange, New Jersey
  - Comprehensive Epilepsy Center, NYU Medical Center, 403 E. 34th Street, 4th Floor, New York, New York
  - Gertrude H. Sergievsky Center, Columbia University, 630 West 168th Street, P&S Box 16 (no patient enrollment), New York, New York
  - Albert Einstein College of Medicine, 111 East 210th St., The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, 3333 Burnet Avenue, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, 34th and Civic Center Blvd., 6th Floor Wood Bldg-Neurology, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Hospital General Agudos Jose Maria Ramos Mejia, Buenos Aires, Argentina
- University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Weisenberg JLZ, Fitzgerald RT, Constantino JN, Winawer MR, Thio LL; EPGP Investigators. Familial aggregation of status epilepticus in generalized and focal epilepsies. Neurology. 2020 Oct 13;95(15):e2140-e2149. doi: 10.1212/WNL.0000000000010708. Epub 2020 Sep 11. PMID 32917807